CLINICAL TRIAL: NCT07073976
Title: Evaluation of Right Ventricular Function to Predict Weaning Success in the Intensive Care Unit: A Prospective Observational Study
Brief Title: Evaluation of Right Ventricular Function to Predict Weaning Success in the Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Weaning-Right Heart
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Weaning Failure of Mechanical Ventilation
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically Ventilated ICU Patients Undergoing Weaning: Adult patients receiving mechanical ventilation in the intensive care unit (ICU) who meet clinical criteria for planned weaning and extubation. All patients will undergo bedside transthoracic echocardiography (TTE) to assess right ventricular function prior to extubation.
  Interventions: Diagnostic Test: Transthoracic Echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography (TTE) — Non-invasive ultrasound imaging of the heart to evaluate right ventricular and right atrial function using parameters such as TAPSE, tricuspid S', RV-FAC, right atrial area, and pulmonary valve acceleration time. TTE will be performed once within 2 hours prior to extubation decision as part of routine care.

SUMMARY:
The goal of this prospective observational study is to evaluate whether right ventricular (RV) function parameters assessed via transthoracic echocardiography (TTE) can predict weaning success in adult intensive care unit (ICU) patients who are mechanically ventilated. The main questions it aims to answer are:

Can the TAPSE (Tricuspid Annular Plane Systolic Excursion) value predict successful extubation?

Do other right heart parameters (tricuspid S', RV-FAC, right atrial area, pulmonary valve acceleration time) provide additional prognostic value for weaning outcomes?

Participants will:

Be adult ICU patients planned for weaning from mechanical ventilation.

Undergo transthoracic echocardiography within 2 hours after meeting clinical weaning criteria.

Have the following echocardiographic parameters measured: TAPSE, tricuspid S', RV-FAC, right atrial area, and pulmonary valve acceleration time.

Be monitored for 24 hours after extubation to assess weaning success (defined as no need for reintubation, non-invasive ventilation, or high-flow oxygen support).

DETAILED DESCRIPTION:
This is a prospective, observational, single-center study designed to investigate whether transthoracic echocardiographic (TTE) assessment of right ventricular function can predict weaning success in mechanically ventilated adult ICU patients. The primary objective is to determine the prognostic value of TAPSE (Tricuspid Annular Plane Systolic Excursion) in forecasting successful extubation.

Secondary objectives include the evaluation of additional echocardiographic parameters such as tricuspid annular systolic velocity (S'), right ventricular fractional area change (RV-FAC), right atrial area, and pulmonary valve acceleration time (PVAT). These parameters will be measured via bedside TTE within 2 hours after patients meet clinical weaning criteria and are hemodynamically stable.

All participants will be monitored for 24 hours after extubation. Weaning success is defined as the ability to sustain spontaneous breathing without the need for reintubation, non-invasive ventilation, or high-flow oxygen therapy during this period.

Data collection will include:

Echocardiographic measurements: TAPSE, tricuspid S', RV-FAC, right atrial area, and PVAT.

Demographic and clinical data: age, sex, BMI, ICU admission diagnosis, APACHE II and SOFA scores, ventilation settings, and duration of mechanical ventilation.

Post-extubation follow-up: reintubation, non-invasive ventilation or high-flow oxygen use, SpO₂ values, blood gas analysis, and vital signs.

This study does not involve any interventions beyond standard care. Echocardiography is routinely performed in ICU settings and poses no additional risk to participants.

The results may support the integration of right heart function assessment into routine ICU weaning protocols and improve clinical decision-making by reducing the incidence of weaning failure and associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Receiving invasive mechanical ventilation in the ICU
* Planned extubation (weaning) according to standard clinical criteria
* Hemodynamically stable at the time of transthoracic echocardiography (TTE)
* Ability to undergo echocardiographic assessment within 2 hours prior to extubation
* Informed consent obtained from patient or legal representative

Exclusion Criteria:

* Known severe tricuspid valve disease or congenital heart disease
* Moderate to severe pericardial effusion or cardiac tamponade
* Inadequate acoustic window for transthoracic echocardiography
* Patients requiring urgent or unplanned extubation
* Use of extracorporeal life support (e.g., ECMO) at the time of assessment
* Known pulmonary embolism or acute cor pulmonale
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are receiving invasive mechanical ventilation in the intensive care unit (ICU) and are scheduled for planned extubation based on standard clinical weaning criteria. All participants must be hemodynamically stable and able to undergo transthoracic echocardiographic assessment prior to extubation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Discriminative Ability of TAPSE for Predicting Weaning Success | Within 24 hours after extubation
  Assessment of the predictive accuracy of TAPSE (Tricuspid Annular Plane Systolic Excursion) in identifying weaning success, defined as no requirement for reintubation, non-invasive ventilation, or high-flow oxygen within 24 hours post-extubation.

SECONDARY OUTCOMES:
Discriminative Ability of RV-FAC in Predicting Weaning Success | Within 24 hours after extubation
  To determine the discriminative performance of right ventricular fractional area change (RV-FAC), measured by transthoracic echocardiography, in identifying weaning success.
Discriminative Ability of Tricuspid S' Velocity in Predicting Weaning Success | Within 24 hours after extubation
  To evaluate the ability of tricuspid annular systolic velocity (S'), obtained via tissue Doppler imaging, to discriminate between successful and unsuccessful weaning outcomes.
Correlation of Right Atrial Area With Weaning Outcome | Within 24 hours after extubation
  To assess whether right atrial area measured before extubation is associated with weaning success or failure.
Correlation of Pulmonary Valve Acceleration Time with Predicting Weaning Success | Within 24 hours after extubation
  To investigate whether pulmonary valve acceleration time (PVAT), measured via transthoracic echocardiography, is associated with weaning success.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)